CLINICAL TRIAL: NCT05045417
Title: IL17 in Systemic Lupus Erythematosus Patients: Association With Disease Activity and Organ Damage
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aya Mohamed Ali, Assistant lecturer of rheumatology and rehabilitation sohag university hospitals, Sohag University
Other Study IDs: Soh-Med-21-09-22
Record Dates: First submitted 2021-09-12; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases with SLE: 110 patients with SLE will be divided to :
  * 40 patients with lupus nephritis
  * 40 patients interstitial lung disease
  * 30 SLE patients without internal organ affection)
  Interventions: Diagnostic Test: Serum level of IL-17
- control group: 30 sex and age matched healthy individuals as a control group
  Interventions: Diagnostic Test: Serum level of IL-17

INTERVENTIONS:
Diagnostic Test: Serum level of IL-17 — Measurement of serum level of IL-17 :
  1. To explore the role of IL-17 in systemic lupus erythematosus
  2. To determine the relation between IL-17 and lupus disease activity
  3. To analyze the correlation between IL-17 and internal organ affection (lupus nephritis , interstitial lung disease)

SUMMARY:
Many laboratory markers can be measured for assessment of Lupus activity as aberrant manufacturing and imbalance of the cytokines of T-helper cell which already have been implicated within autoimmunity pathogenesis as IL-18 and IL-10 levels are usually elevated in lupus sufferers and correlated with SLEDAI score IL-17 has been linked to immune-mediated organ damage in several autoimmune diseases and recently it has been linked to pathogenesis of a murine model of lupus and human lupus Diverse cytokine abnormalities which common in lupus patients may skew T cells differentiation into IL-17-producing CD4+ and double negative T cells. This could promote the autoimmune process by activation of immune cells &stimulation of proliferation of B-cell and production of antibody

ELIGIBILITY:
Inclusion Criteria:

* SLE will be diagnosed according to the 2012 Systemic Lupus International Collaborating Clinics (SLICC) classification criteria for SLE
* Age ≥ 18 years.
* Patients who are able and willing to give written informed consent

Exclusion Criteria:

-Any other autoimmune disease rather than SLE. -

* Systemic diseases
* Malignancy
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * The study will include 110 patients with SLE :
    * 40 with lupus nephritis
    * 40 with interstitial lung disease
    * 30 SLE patients without internal organ affection)
  * In addition to 30 sex and age matched healthy individuals as a control group
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
SLE disease activity index (SLEDAI) | 18 Months
  • Assessment of the disease activity in the patients will be done by using the SLE disease activity index (SLEDAI). It potentially measures reversible manifestations of the underlying inflammatory disease process. The scale includes24 "weighted" attribute grouped into 9 domains. The final score is the sum of all attributed scores.
  * No activity 0
  * mild activity: 1-5
  * moderate activity: 6- 1 0
  * high activity : 1 1 - 1 9
  * very high > 20

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Crispin JC, Tsokos GC. IL-17 in systemic lupus erythematosus. J Biomed Biotechnol. 2010;2010:943254. doi: 10.1155/2010/943254. Epub 2010 Apr 6. PMID 20379379
- [Background] Garrett-Sinha LA, John S, Gaffen SL. IL-17 and the Th17 lineage in systemic lupus erythematosus. Curr Opin Rheumatol. 2008 Sep;20(5):519-25. doi: 10.1097/BOR.0b013e328304b6b5. PMID 18698171
- [Background] Su DL, Lu ZM, Shen MN, Li X, Sun LY. Roles of pro- and anti-inflammatory cytokines in the pathogenesis of SLE. J Biomed Biotechnol. 2012;2012:347141. doi: 10.1155/2012/347141. Epub 2012 Feb 15. PMID 22500087